CLINICAL TRIAL: NCT02248701
Title: Higher-Than-Replacement Testosterone Plus Finasteride Treatment After SCI
Brief Title: Testosterone Plus Finasteride Treatment After Spinal Cord Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment difficulties
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B1449-R; 1I01RX001449-01A1 (NIH)
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Spinal Cord Injury; Spinal Cord Injuries; Trauma, Nervous System; Wounds and Injuries; Central Nervous System Diseases; Nervous System Diseases; Spinal Cord Diseases; Gonadal Disorders; Endocrine System Diseases; Hypogonadism; Genital Diseases, Male
Keywords: Testosterone; Testosterone enanthate; Testosterone undecanoate; Testosterone 17 beta-cypionate; Methyltestosterone; Androgens; Hormones; Hormone Substitutes, and Hormone Antagonists; Physiologic Effects of Drugs; Pharmacologic Actions; Antineoplastic Agents, Hormonal; Antineoplastic Agents; Therapeutic Uses; Anabolic Agents; Testosterone Replacement Therapy; Dual Energy X ray Absorptiometry; Lean Tissue Mass; Body Composition; Lipid and Glucose profile; Muscle Strength; 5-alpha Reductase; Muscle Mass; Bone Mineral Density; Adipose Tissue; Body Fat; Density, Bone; Bone Formation; Bone Resorption; Bone Density Conservation Agents; Magnetic Resonance Imaging; Muscle, Skeletal; Bone and Bones; Gait; Walking; Locomotion; Motor Activity
MeSH Terms: conditions — Spinal Cord Injuries; Trauma, Nervous System; Wounds and Injuries; Central Nervous System Diseases; Nervous System Diseases; Spinal Cord Diseases; Gonadal Disorders; Endocrine System Diseases; Hypogonadism; Genital Diseases, Male; Bone Resorption; Motor Activity | interventions — testosterone enanthate; Finasteride; Sesame Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- testosterone enanthate, finasteride (Experimental): Testosterone enanthate via i.m. injection (125 mg/week) and finasteride orally (5 mg/day)
  Interventions: Drug: Testosterone Enanthate; Drug: Finasteride
- placebo treatment (Placebo Comparator): Placebo via i.m. injection (once weekly) and placebo pill orally (daily)
  Interventions: Drug: Placebo injection; Drug: Placebo pill

INTERVENTIONS:
Drug: Testosterone Enanthate — Subjects receive testosterone (125 mg/week) by intramuscular injection
  Other Names: delatestryl
  Arms: testosterone enanthate, finasteride
Drug: Finasteride — Subjects receive finasteride (5 mg/day) orally
  Other Names: proscar
  Arms: testosterone enanthate, finasteride
Drug: Placebo injection — Subjects receive placebo (weekly) by intramuscular injection
  Other Names: sesame oil
  Arms: placebo treatment
Drug: Placebo pill — Subjects receive placebo pill (daily) orally
  Other Names: inactive substance
  Arms: placebo treatment

SUMMARY:
The purpose of this study is to determine whether testosterone plus finasteride treatment will improve musculoskeletal health, neuromuscular function, body composition, and metabolic health in hypogonadal men who have experienced ambulatory dysfunction subsequent to incomplete spinal cord injury. The investigators hypothesize that this treatment will improve bone mineral density, enhance muscle size and muscle function, and improve body composition, without causing prostate enlargement.

DETAILED DESCRIPTION:
Men with spinal cord injury (SCI) experience a high prevalence of hypogonadism which influences the neural, muscular, skeletal, and body composition deficits that occur after injury. It remains unknown whether testosterone administration improves bone mineral density, muscle mass and muscle function, and body composition / metabolic health in hypogonadal men who have experienced ambulatory dysfunction subsequent to incomplete spinal cord injury. In addition, it is unknown whether testosterone or the 5-alpha reduced metabolite dihydrotestosterone (an endogenous metabolite of testosterone) mediate effects in these and other tissues.

For this study hypogonadal men with motor incomplete spinal cord injury who present with ambulatory dysfunction will be randomized to receive testosterone plus the 5-alpha reductase inhibitor finasteride or a placebo treatment for 12 months. Testosterone or placebo injection will be administered weekly; finasteride or placebo will be administered daily. Participants will be assessed at study entry and at 1-6 month intervals thereafter. Assessments will include measurements such as a dual energy x-ray absorptiometry (DEXA) scan, MRI scan, and muscle performance tests. Participants will also have several safety tests, including electrocardiogram (EKG) for cardiac electrophysiology, prostate digital rectal exam and prostate ultrasound sizing for prostate health, and blood tests to assess hematocrit, liver enzymes (AST and ALT), prostate specific antigen (PSA), cholesterol, and other health markers.

ELIGIBILITY:
Inclusion Criteria:

* Male > 18 years of age
* Traumatic, vascular, or orthopedic spinal cord injury between C2-L3 >12 months prior to enrollment
* Motor incomplete spinal cord (AIS C/D)
* Ambulatory dysfunction
* Medically stable condition that is asymptomatic for bladder infection, decubiti, cardiopulmonary disease, or other significant medical conditions
* Serum total testosterone (<325 ng/dL) or bioavailable testosterone (<70 ng/dL)

Exclusion Criteria:

* Currently participating in another research protocol that may influence study outcomes
* Life expectancy <1 year
* History of or current congenital spinal cord injury or other degenerative spinal disorder
* Diagnosis of multiple sclerosis, amyotrophic lateral sclerosis, or other neurologic impairment/injury
* History of venous thromboembolism within the last 6 months, specifically deep venous thromboembolism and pulmonary embolism, history of recurrent venous thromboembolism or know hereditary thrombophilia
* Poorly compensated or uncontrolled cardiovascular disease
* Any major cardiovascular event within the last 12 months (defined as a history of acute myocardial infarction, any cardiac revascularization procedure including angioplasty, stenting, or coronary artery bypass grafting, hospitalization due to unstable angina, transient ischemic attack, or stroke)
* Any angina that is not controlled on a current medical regimen (Canadian class II, III, or IV)
* New York Heart Association (NYHA) class III or IV congestive heart failure
* Systolic blood pressure >160 mmHg or diastolic blood pressure >100 mm Hg
* Poorly controlled arrhythmia
* Severe valvular disease
* LDL cholesterol >160 mg/dl with known history of any major cardiovascular event, as defined above, within the last 12 months
* Baseline EKG findings (e.g. left bundle branch block) or marked EKG abnormalities that would preclude serial screening for occult ischemic events
* Current prostate, breast, or other organ cancer
* History of prostate, breast, or other organ cancer, with the exceptions of completely resolved basal or squamous cell carcinoma for a duration of >24 months or completely resolved melanoma for a duration of >24 months
* Serum prostate-specific antigen (PSA) >3.0 ng/ml
* History of benign prostate enlargement (BPE) >40cc, evaluated via TRUS
* Hematocrit >47%
* Liver enzymes (AST / ALT) above normal upper limit
* Creatinine >1.4 mg/dL
* Serum calcium >10.5 mg/dL
* Gynecomastia
* Mental state that precludes understanding of the protocol
* Diagnosed, but untreated moderate or severe sleep apnea
* Spinal nutrition screening tool score >15
* Severe claustrophobia that precludes MRI testing
* Current anticoagulant therapy
* Use of any of the following pharmacologic agents in the previous 3 months (testosterone, leuprolide, androgenic hormones, growth hormone, oral androgen precursors, 5-alpha reductase or aromatase inhibitors)
* Use of anti-resorptive or bone anabolic drug therapy in the previous 6 months
* Known allergy to sesame oil

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be male
Enrollment: 33 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua F Yarrow, PhD MS BS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL; Dana M Otzel, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (2):
- United States (2):
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to the requirements described by the Department of Veterans Affairs, Office of Research & Development.
Time Frame: Data will be shared according to the requirements described by the Department of Veterans Affairs, Office of Research & Development.
Access Criteria: Data will be shared according to the requirements described by the Department of Veterans Affairs, Office of Research & Development.

REFERENCES:
- [Derived] Otzel DM, Nichols L, Conover CF, Marangi SA, Kura JR, Iannaccone DK, Clark DJ, Gregory CM, Sonntag CF, Wokhlu A, Ghayee HK, McPhaul MJ, Levy CE, Plumlee CA, Sammel RB, White KT, Yarrow JF. Musculoskeletal and body composition response to high-dose testosterone with finasteride after chronic incomplete spinal cord injury-a randomized, double-blind, and placebo-controlled pilot study. Front Neurol. 2024 Dec 11;15:1479264. doi: 10.3389/fneur.2024.1479264. eCollection 2024. PMID 39722695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referrals at 2 VA medical centers and via community-based advertisements between January 2017 and March 2021 and pre-screened via phone to determine criteria to enroll. Those meeting criteria to enroll were screened for potential eligibility, with the first participant enrolled on April 27, 2017 and the last participant enrolled on December 4, 2020.
Pre-assignment Details: Enrolled participants were evaluated at an in-person screening visit to determine if they qualify. Those that did not qualify were excluded from the study before randomization. Of 33 enrolled participants, 12 met inclusion criteria and were randomized to treatment / placebo groups.
Period: Overall Study
Arm/Group | Testosterone Enanthate, Finasteride | Placebo Treatment
Started | 7 | 5
Completed | 3 | 3
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — VA mandated stop on all in person visits for VA sponsored research nationally | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Enanthate, Finasteride | Placebo Treatment | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (6.3) | 57.4 (9.4) | 60.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12
Hip bone mineral density [Mean (Standard Deviation); unit: g/cm^2] — non-dominant leg total hip bone mineral density, assessed via DXA Population: N=1 participant in the was not analyzed in the testosterone enanthate, finasteride group due to bilateral hip joint replacement present at baseline.
  g/cm^2
    number analyzed (Participants) | 6 | 5 | 11
    (all) | 0.9788 (0.2073) | 1.016 (0.1365) | 0.996 (0.1712)
Thigh muscle cross-sectional area [Mean (Standard Deviation); unit: cm^2] — non-dominant leg knee extensors muscle cross-sectional area, assessed via MRI
  cm^2 | 7483 (2096) | 6453 (1177) | 7054 (1783)
Total body fat [Mean (Standard Deviation); unit: kg] — assessed via DXA Population: Only N=6 analyzed in the testosterone enanthate, finasteride group because data was corrupted at baseline on N=1 participant.
  kg
    number analyzed (Participants) | 6 | 5 | 11
    (all) | 30.4 (8.7) | 30.3 (9.6) | 30.3 (8.6)
Walking speed [Mean (Standard Deviation); unit: m/s] — assessed via 10m walking test
  m/s | 0.90 (0.33) | 0.76 (0.35) | 0.84 (0.33)
Neuromuscular function [Mean (Standard Deviation); unit: N/m] — non-dominant leg, thigh (knee extensors) peak isometric torque production via dynamometry
  N/m | 121 (37) | 111 (36) | 117 (35)
Visceral fat [Mean (Standard Deviation); unit: kg] — Android fat assessed via DXA Population: Only N=6 analyzed in the testosterone enanthate, finasteride group because data was corrupted at baseline on N=1 participant.
  kg
    number analyzed (Participants) | 6 | 5 | 11
    (all) | 2.85 (1.00) | 3.19 (1.61) | 3.00 (1.25)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Hip Bone Mineral Density
Description: Percent change in total hip bone mineral density of the non-dominant limb assessed via dual-energy X-ray absorptiometry (DXA)
Time Frame: Baseline, 6 months, 12 months
Population: Only 5 participants in the testosterone enanthate group were evaluated because 1 of 6 with baseline values had withdrawn prior to 6 months. At 12 months: 2 participants in the placebo group and 2 additional participants in the testosterone enanthate group had withdrawn from the study and data from 1 participant in the testosterone enanthate group could not be analyzed due to imaging artefact.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Testosterone Enanthate, Finasteride | Placebo Treatment
Number analyzed (Participants) | 5 | 5
percent change
  Change at 6 months | 1.7 (4.7) | -0.5 (2.4)
  Change at 12 months: number analyzed (Participants) | 2 | 3
  Change at 12 months | 1.2 (7.3) | 1.1 (4.9)

2. Primary Outcome: Percent Changes in Muscle Cross-Sectional Area
Description: Percent Change in thigh (knee extensors) muscle cross-sectional area of the non-dominant limb assessed via MRI
Time Frame: Baseline, 6 months, 12 months
Population: Only 5 participants in the testosterone enanthate group were evaluated because 2 of 7 with baseline values had withdrawn prior to 6 months. Only 4 participants in the placebo group were evaluated because 1 of 5 with baseline values did not have a follow-up MRI. At 12 months: 1 participant in the placebo group and 2 additional participants in the testosterone enanthate group had withdrawn from the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Testosterone Enanthate, Finasteride | Placebo Treatment
Number analyzed (Participants) | 5 | 4
percent change
  6 months | 7.9 (4.4) | -0.9 (4.1)
  12 months: number analyzed (Participants) | 3 | 3
  12 months | 11.4 (6.0) | -1.9 (4.3)

3. Primary Outcome: Percent Change in Total Body Fat
Description: Percent change in total body fat assessed via dual-energy x-ray absorptiometry (DXA)
Time Frame: Baseline, 6 months, 12 months
Population: Only 4 participants in the testosterone enanthate group were evaluated because 2 of 6 with baseline values had withdrawn prior to 6 months. At 12 months: 2 participants in the placebo group had withdrawn from the study and 2 additional participants in the testosterone enanthate group had withdrawn from the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Testosterone Enanthate, Finasteride | Placebo Treatment
Number analyzed (Participants) | 4 | 5
percent change
  6 months | -6.8 (5.0) | -4.7 (10.6)
  12 months: number analyzed (Participants) | 2 | 3
  12 months | -8.7 (8.4) | -1.9 (9.1)

4. Primary Outcome: Absolute Change in Walking Speed
Description: Absolute change in 10 m walking speed
Time Frame: Baseline, 6 months, 12 months
Population: Only 5 participants in the testosterone enanthate group were evaluated because 2 of 7 with baseline values had withdrawn prior to 6 months. At 12 months: 2 participants had withdrawn from the placebo group and an additional 2 participants had withdrawn from the testosterone enanthate group.
Measure: Mean (Standard Deviation); unit: meters/second (m/s) change
Arm/Group | Testosterone Enanthate, Finasteride | Placebo Treatment
Number analyzed (Participants) | 5 | 5
meters/second (m/s) change
  6 months | 0 (0.17) | 0.05 (0.14)
  12 months: number analyzed (Participants) | 3 | 3
  12 months | 0.10 (0.12) | 0.01 (0.15)

5. Secondary Outcome: Percent Change in Neuromuscular Function
Description: Percent change in thigh (knee extensors) peak isometric torque production of the non-dominant limb assessed via dynamometry
Time Frame: Baseline, 6 months, 12 months
Population: Only 5 participants in the testosterone enanthate group were evaluated because 2 of 7 with baseline values had withdrawn prior to 6 months. At 6 months: 1 participant in the placebo group and 1 participant in the testosterone enanthate group did not perform testing. At 12 months: 2 participants in the placebo group had withdrawn from the study and 2 additional participant in the testosterone enanthate group had withdrawn from the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Testosterone Enanthate, Finasteride | Placebo Treatment
Number analyzed (Participants) | 5 | 5
percent change
  6 months: number analyzed (Participants) | 4 | 4
  6 months | 19.9 (30.7) | -8.6 (14.9)
  12 months: number analyzed (Participants) | 3 | 3
  12 months | 15.5 (27.0) | 0.5 (35.1)

6. Secondary Outcome: Percent Change in Visceral Fat
Description: Percent change in visceral (android) fat mass assessed via dual-energy x-ray absorptiometry (DXA)
Time Frame: Baseline, 6 months, 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Testosterone Enanthate, Finasteride | Placebo Treatment
Number analyzed (Participants) | 4 | 5
percent change
  6 months | -8.2 (17.0) | -3.2 (7.7)
  12 months: number analyzed (Participants) | 2 | 3
  12 months | -13.6 (9.4) | 0.2 (11.6)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Data on adverse events were assessed at regular study visits and via weekly phone assessments with all study participants.
Arm/Group | Testosterone Enanthate, Finasteride | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/5
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Enanthate, Finasteride (N=7) | Placebo Treatment (N=5)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0) — Hospitalization due to severe acute respiratory syndrome (SARS)-CoV-2 (COVID-19) infection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Enanthate, Finasteride (N=7) | Placebo Treatment (N=5)
aldolase, high (General disorders) | 1 (1) | 0 (0) — above standard reference range (<=8.1 U/L); test performed on only 1 participant at request of study physician
anion gap, high (General disorders) | 1 (1) | 2 (3) — above standard reference range (5-15 mmol/L)
alanine aminotransferase (ALT), high (Investigations) | 2 (2) | 1 (1) — above standard reference range (0-40 U/L)
aspartate aminotransferase (AST), high (Investigations) | 1 (1) | 0 (0) — above standard reference range (0-45 U/L)
albumin, high (General disorders) | 0 (0) | 1 (1) — above standard reference range (3.5-5.0 g/dL)
alkaline phosphatase, high (General disorders) | 0 (0) | 1 (4) — above standard reference range (0-125 U/L)
calcium, high (Investigations) | 1 (2) | 1 (1) — above standard reference range (8.4-10.5 mg/dL)
total cholesterol, high (Investigations) | 4 (14) | 2 (5) — above standard reference range (0-199 mg/dL); all participants in testosterone enanthate, finasteride group exhibited cholesterol values above standard reference range at baseline (before treatment initiation)
chloride, low (General disorders) | 0 (0) | 1 (1) — below standard reference range (98-108 mmol/L)
CO2, low (General disorders) | 2 (7) | 1 (1) — below standard reference range (23-32 mmol/L)
creatine phosphokinase (CPK), high (General disorders) | 1 (2) | 0 (0) — above standard reference range (5-180 U/L); test performed on only 1 participant at request of study physician
creatinine, high (General disorders) | 2 (3) | 2 (2) — above standard reference range (0.5-1.2 mg/dL)
C-reactive protein (CRP), high (General disorders) | 6 (18) | 3 (9) — above standard reference range (<0.1-0.4 mg/dL); 3 of 6 testosterone enanthate, finasteride participants and 1 of 3 placebo participants with elevated CRP exhibited values above standard reference range at baseline (before treatment initiation)
dihydrotestosterone, high (Investigations) | 0 (0) | 1 (2) — above standard reference range (16-79 ng/dL)
dihydrotestosterone, low (Investigations) | 5 (13) | 2 (8) — below standard reference range (16-79 ng/dL)
dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
edema (Investigations) | 1 (2) | 0 (0) — present in upper and lower extremities
impaired ejaculation (Reproductive system and breast disorders) | 0 (0) | 1 (2) — patient reported outcome
estradiol, high (Investigations) | 7 (28) | 4 (7) — above standard reference range (<=29 pg/mL)
eosinophils, high (General disorders) | 5 (22) | 5 (12) — above standard reference range (0-3%)
erythropoietin, high (General disorders) | 2 (9) | 2 (5) — above standard reference range (2.6-18.5 mIU/mL)
eye infection (Eye disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 1 (1) | 0 (0) — transient depression, self reported
falls (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
glucose, high (Investigations) | 7 (29) | 5 (23) — above standard reference range (65-99 mg/dL); 7 of 7 participants in testosterone enanthate, finasteride group and 3 of 5 participants in placebo group exhibited glucose values above standard reference range at baseline (before treatment initiation)
granulocytes, high (General disorders) | 1 (4) | 4 (12) — above standard reference range (54-65%)
granulocytes, low (General disorders) | 4 (11) | 3 (8) — below standard reference range (54-65%)
HDL cholesterol, low (Investigations) | 5 (14) | 2 (13) — below standard reference range (>=40 mg/dL); 3 of 5 participants in testosterone enanthate, finasteride group and 2 of 2 participants in placebo group with low HDL exhibited values below reference range at baseline (before treatment initiation)
hematocrit, high (Investigations) | 0 (0) | 1 (1) — above standard reference range (41-52%)
hematocrit, low (Investigations) | 1 (4) | 3 (17) — below standard reference range (41-52%)
hemoglobin, high (Investigations) | 0 (0) | 1 (1) — above standard reference range (13.9-18 g/dL)
hemoglobin, low (Investigations) | 2 (9) | 3 (15) — below standard reference range (13.9-18 g/dL)
insulin, high (Investigations) | 2 (2) | 4 (20) — above standard reference range (<=19.6 uIU/mL)
potassium, high (General disorders) | 1 (1) | 0 (0) — above standard reference range (3.5-5.0 mmol/L)
potassium, low (General disorders) | 0 (0) | 2 (2) — below standard reference range (3.5-5.0 mmol/L)
LDL cholesterol, high (Investigations) | 3 (12) | 0 (0) — above standard reference range (<=129 mg/dL); 3 of 3 participants in testosterone enanthate, finasteride group with high LDL cholesterol exhibited values above standard reference range at baseline (before treatment initiation)
lymphocytes, high (General disorders) | 3 (7) | 2 (6) — above standard reference range (25-33%)
lymphocytes, low (General disorders) | 3 (11) | 4 (17) — below standard reference range (25-33%)
mean corpuscular hemoglobin, low (General disorders) | 2 (7) | 0 (0) — below standard reference range (27-33.3 pg)
mean corpuscular hemoglobin concentration, low (General disorders) | 3 (8) | 1 (1) — below standard reference range (31.8-37.1 g/dL)
mean corpuscle volume, high (General disorders) | 0 (0) | 1 (1) — above standard reference range (80-98 um^3)
mean corpuscle volume, low (General disorders) | 1 (5) | 0 (0) — below standard reference range (80-98 um^3)
monocytes, high (General disorders) | 7 (34) | 5 (23) — above standard reference range (3-7%); 6 of 7 participants in testosterone enanthate, finasteride group and 3 of 5 participants in placebo group exhibited monocyte values above standard reference range at baseline (before treatment initiation)
mean platelet volume, high (General disorders) | 4 (5) | 3 (5) — above standard reference range (7.4-10.5 um^3)
myelocytes, high (General disorders) | 1 (1) | 0 (0) — above standard reference range (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (5) — self reported
otitis media (Ear and labyrinth disorders) | 1 (1) | 0 (0) — ear infection
paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
penile shrinkage (Reproductive system and breast disorders) | 1 (1) | 0 (0) — self reported
total protein, high (General disorders) | 1 (1) | 1 (1) — above standard reference range (6.0-8.2 g/dL)
prostate-specific antigen (PSA), high (Investigations) | 2 (3) | 0 (0) — above standard reference range (0-4 ng/mL or increase >1.4 ng/mL vs baseline); 1 of 2 participants in testosterone enanthate, finasteride group with high PSA tested positive for urinary tract infection 2 different times with PSA renormalizing
prostate induration (Investigations) | 0 (0) | 1 (1) — noted on digital rectal exam of prostate
red blood cell count, low (General disorders) | 2 (3) | 3 (12) — below standard reference range (4.44-6.1 M/cmm)
red blood cell distribution width, high (General disorders) | 3 (9) | 0 (0) — above standard reference range (39.0-52.2 fL)
red blood cell distribution width, low (General disorders) | 0 (0) | 2 (6) — below standard reference range (39.0-52.2 fL)
segmented neurtrophils, low (General disorders) | 1 (1) | 0 (0) — below standard reference range (54-65%)
sex-hormone binding globulin (SHBG), high (General disorders) | 0 (0) | 1 (3) — above standard reference range (10-50 nmol/L)
sex-hormone binding globulin (SHBG), low (General disorders) | 0 (0) | 1 (5) — below standard reference range (10-50 nmol/L)
sodium, high (General disorders) | 0 (0) | 1 (1) — above standard reference range (135-145 mmol/L)
testicular size reduced (Reproductive system and breast disorders) | 1 (1) | 0 (0) — self reported outcome
testosterone, high (Investigations) | 5 (12) | 0 (0) — above standard reference range (193-836 ng/dL)
testosterone, low (Investigations) | 2 (2) | 1 (7) — below standard reference range (193-836 ng/dL)
triglycerides, high (Investigations) | 4 (11) | 3 (17) — above standard reference range (0-149 mg/dL)
urea nitrogen, high (General disorders) | 0 (0) | 2 (2) — above standard reference range (9-20 mg/dL)
urea nitrogen, low (General disorders) | 2 (4) | 0 (0) — below standard reference range (9-20 mg/dL)
urobilinogen, high (General disorders) | 1 (1) | 0 (0) — above standard reference range (0.00-1.99 mg/dL)
urinary tract infection (Renal and urinary disorders) | 1 (2) | 0 (0) — As a result of self-catheterization
white blood cell count, high (General disorders) | 1 (1) | 1 (1) — above standard reference range (4.6-10.8 k/cmm)
white blood cell count, low (General disorders) | 1 (1) | 0 (0) — below standard reference range (4.6-10.8 k/cmm)

LIMITATIONS AND CAVEATS:
This trial was terminated early due to enrollment and retention difficulties that persisted during the severe acute respiratory syndrome (SARS)-Cov19 pandemic. This resulted in a smaller number of subjects being enrolled and undergoing testing than was originally planned in our a priori analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT02248701/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT02248701/ICF_001.pdf